



City Hospital Dudley Road Birmingham B18 7QH

Tel: 0121 554 3801 www.swbh.nhs.uk

## **CONSENT FORM**

| Patient Identification Number: | | | | |
|---|---|---|---|---|
| Name of the Researcher: | | | | |
| Study: | CT coronary angiogram percutaneous coronary a | | | cked artery (CTO) |
| 1. I confirm that I have read and understood the patient information sheet version 1 dated 28/02/2021 for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | | |
| | | | Please initial box: | |
| | stand that my participation is<br>giving any reason, and that | | | |
| | | | Please initial box: | |
| 3. I understand that relevant sections of my medical notes/study data may be looked at by responsible individuals from the Study Team, the Sponsor, NHS Trust or by Regulatory Bodies, where it is relevant to my taking part in this research. I give permission for these individuals to access my records. | | | | |
| | | | Please initial box: | |
| 4. I agree for my GP to be informed of my participation in the study. | | | | |
| | | | Please initial box: | |
| 5. I agree to take part in the above study. | | | | |
| | | | Please initial box: | |
| 6. I agree for one set of blood samples to be drawn for routine tests | | | | |
| | | | Please initial box: | |
| Name of p | patient | Date | Signature | |
| Name of I | Researcher | Date | Signature | |



City Hospital Dudley Road Birmingham B18 7QH

Tel: 0121 554 3801 www.swbh.nhs.uk

Was a Trust interpreter used to translate the patient information sheet and take consent?: Yes/No (please circle as appropriate)

Signature of the interpreter below to confirm that the study details from the patient information sheet was accurately translated and all questions answered satisfactorily:

| Name of Interpreter | /Language | Date | Signature |
|---|---|---|---|
| Witness (Name) | | Date | Signature |
| Results of the study | | | |
| Would you like results of the study to be mailed to you: Yes/No (circle appropriate) (If yes, mailing address to be kept separately) | | | |
| When completed: | 1 copy in care 1 copy for part 1 copy for rese | ticipant | |